CLINICAL TRIAL: NCT03529292
Title: Pilot Study to Evaluate the Safety and the Efficacy of the Filling Using the Matrix and Cells, Obtained by the AmeaCell® Device From Autologous Adipose Tissue and Intended for the Filling of Wrinkles on the Face.
Brief Title: Pilot Study to Evaluate the Safety and the Efficacy of the Matrix and Cells Obtained by the AmeaCell® Device and Intended for the Filling of Wrinkles on the Face.
Acronym: SKINMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Symbioken (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYMB-SAF1701
Record Dates: First submitted 2018-05-04; First posted 2018-05-18 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Skin Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Matrix and Cells obtained by the AmeaCell® device (Experimental)
  Interventions: Device: AmeaCell

INTERVENTIONS:
Device: AmeaCell — Lipoaspirate obtained from liposuction is treated by the AmeaCell® device in order to obtain Matrix and Cells which contains cellular phase and matrix phase. The Matrix ancd Cells are injected in the same patient as facial wrinkles filler.

SUMMARY:
The purpose of this study is to evaluate the filling using the Matrix and Cells, obtained by the Ameacell® device from autologous adipose tissue and intended for the filling of wrinkles on the face.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the filling using the Matrix and Cells, obtained by the Ameacell® device from autologous adipose tissue and intended for the filling of wrinkles on the face.

This is a mono-center, pilot study in 24 subjects

ELIGIBILITY:
Inclusion Criteria:

* Man or woman from 18 to 70 years
* Subject wishing liposuction
* Subject wishing a filling of facial wrinkles for aesthetic purposes
* Subject for which it is possible to achieve a puncture of adipose tissue of at least 150ml so that after decantation or centrifugation there remains 100ml of adipose tissue
* Facial wrinkles that can be treated with the Matrix and Cells volume of approximately 12ml
* Grade of wrinkles at level 2 minimum of the nasolabial fold according to the WSRS scale
* Free, informed and written consent
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Pregnant or breastfeeding woman or planning to be pregnant
* Woman of childbearing age without effective contraceptive
* Subject having a filling of facial wrinkles with hyaluronic acid or by a method of lipofilling (injection of adipose tissue) in the 12 months prior to the enrollment
* Subject who has undergone treatment of facial wrinkles by injection of botulinum toxin, by mesotherapy or cosmetic procedure (laser, photo modulation, intense pulsed light, radio frequency, dermabrasion, chemical peel or other ablative procedures) within 12 months at least prior to enrolment or subject who is planning this type of procedure during the study
* Subject who has received semi-permanent dermal fillers or permanent facial implants or who is planning to do this type of implant during the study
* Subject having history of formation of hypertrophic scars or keloids
* Subject having a skin disease or skin inflammation (e.g. acne, herpes, eczema, psoriasis, sclerosis) at the site to be treated or elsewhere on the body if suspected of spreading on the site to be treated
* Subject with allergic contact dermatitis or a history of allergic contact dermatitis or a family history of allergic contact dermatitis
* Presence of tattoo and / or scar in the treatment area that, in the opinion of the investigator, could interfere with the evaluation of the study
* Diabetes (type I or type II)
* Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) seropositivity
* Subject under anti-HIV treatment
* Autoimmune disease
* Immunodepression
* History of phlebitis or pulmonary embolism
* Major pathology involving the renal, hepatic, cardiovascular, immune and / or nervous system
* Cancerous lesion on the face
* Any other diseases that could, in the opinion of the investigator, be clinically significant and make the subject inappropriate for the study, alter the results of the study or increase the risk for the subject
* Known hypersensitivity to cobalt
* Known hypersensitivity to collagenase
* Known or suspected allergy to lidocaine or any other amide anesthetic
* History of known severe allergies (anaphylaxis, angioedema) for a product used in the study
* Any contraindication to lipofilling surgery
* Active smoking or subject who stopped smoking less than one month before the intervention
* Radiotherapy treatment at the head and neck region.
* Chemotherapy treatment
* Treatment with anticoagulant or Nonsteroidal anti-inflammatory drug (NSAID) or any other substance known to increase clotting time during the 2 weeks prior to enrollment
* Corticosteroids in the 6 weeks prior to enrollment
* Subject having a metal-metal hip prosthesis
* Subject under lidocaine or structurally related local anesthetic (e.g. bupivacaine) within 24 hours prior to enrollment
* Subject having undergone general anesthesia for less than 8 days
* Treatment with an oral or topical retinoid in the month prior to enrollment
* Subject having a history of drug or alcohol addiction in the 12 months prior to enrollment
* Participation in another research including an exclusion period still in progress at the time of enrollment
* Person placed under guardianship or curatorship or under the protection of justice

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of the Adverse Event(s) | From selection up to 12 months after the injection
  Adverse events will be investigated and recorded at each visit by the investigator
Local tolerance | First 4 weeks after the injection
  The subject will record daily the local tolerance in a diary card. Signs of erythema, edema, bruising, discolouration, pain / tenderness, and pruritus will be noted and scored from 0 (none) to 3 (severe).

SECONDARY OUTCOMES:
Wrinkle Severity Rating Scale (WSRS) Evaluation for the nasolabial folds | Change from baseline at month 1, 6 and 12
  The Wrinkle Severity Rating Scale (WSRS) is a 5-point reference scale with photographs that classifies deep facial wrinkles (Nasolabial Folds). The grading is performed on both sides to give a reliable and reproducible gradation of the depth of the folds. The grading of the wrinkles is made by the investigator according to the following grades:
  Grade 1 No visible nasolabial folds; continuous skin line Grade 2 Shallow but visible nasolabial folds with a slight indentation Grade 3 Moderate deep nasolabial folds; visible at normal appearance Grade 4 Very long and deep nasolabial folds; prominent facial feature ;< 2mm visible fold if stretched Grade 5 Extreme deep long nasolabial folds; 2-4mm V shaped fold if stretched
Depth of the wrinkles by 3D picture | Change from baseline at month 1, 6 and 12
Global Aesthetic Improvement Scale (GAIS) Evaluation | Change from baseline at month 1, 6 and 12
  The GAIS scale ("Global Aesthetic Improvement Scale") is a judgment scale noting the apparent overall aesthetic improvement, in comparison with the aspect observed before the injection (on a photograph taken during the day of inclusion). Rating categories are: "Worse"; "No change"; "Slightly improved", "Much improved"; "Very much improved".
  Evaluations are carried out by the investigator but also by the subject himself according to the same criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Cuylits, Principal Investigator — Hôpital Erasme, Bruxelles, BELGIUM
Locations (1):
- Hôpital Erasme, Brussels, Belgium